CLINICAL TRIAL: NCT01459471
Title: Staple-line Reinforcement During Laparoscopic Sleeve Gastrectomy Using Three Different Techniques: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Gentileschi, Professor, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEND-11-0905
Record Dates: First submitted 2011-10-04; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Complication of Surgical Procedure; Leak; Blood
MeSH Terms: interventions — Bariatric Surgery; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bleeding, leak, operative time (Experimental)
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Staple line reinforcement during sleeve gastrectomy
  Other Names: bariatric surgical procedure; gastric resection; steaple line reinforcement

SUMMARY:
The main drawback of laparoscopic sleeve gastrectomy (LSG) is the severity of post-operative complications. Staple line reinforcement (SLR) is strongly advocated.

DETAILED DESCRIPTION:
The aim of this study was to prospectively and randomly compare three different techniques of SLR during LSG: oversewing (group A), buttressed transection with a polyglycolide acid and trimethylene carbonate (group B) and staple-line roofing with a gelatin fibrin matrix (group C).

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients waiting for sleeve gastrectomy

Exclusion Criteria:

* BMI<35 Kg/m2,
* Important comorbidities

Ages: 28 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
safety of staple line reinforcement during laparoscopic sleeve gastrectomy by measuring the number of adverse effects, i.e. bleeding and leaks. | six months
  a comparison between three techniques of staple line reinforcement. The number of adverse events will be registered and analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gentileschi, MD, Study Director — University of Tor Vergata, Rome, Italy